CLINICAL TRIAL: NCT05326503
Title: Testing a Natural Polyphenol Supplement to Inhibit Dietary Iron Absorption in Thai Adults with Iron-loading Thalassemia: a Stable Isotope Study
Brief Title: Inhibitory Effect of a Polyphenol Supplement on Dietary Iron Absorption in Adults with Thalassemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fe-PP-Thal
Record Dates: First submitted 2022-02-09; First posted 2022-04-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Thalassemia; Iron Overload
Keywords: Iron overload; Thalassemia; Polyphenols; Iron absorption
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Meal with polyphenol supplement (PPS) (Experimental): Iron-rich test meal labelled with stable iron isotope as ferrous sulfate, consumed with the polyphenol supplement.
  Interventions: Dietary Supplement: Meal matrix with polyphenol supplement (PPS)
- Meal with placebo (Placebo Comparator): Iron-rich test meal labelled with stable iron isotope as ferrous sulfate, consumed with placebo supplement (maltodextrin).
  Interventions: Dietary Supplement: Meal matrix with placebo
- Drink with PPS (Experimental): Iron-fortified drink labelled with stable iron isotope as ferrous sulfate, consumed with the polyphenol supplement.
  Interventions: Dietary Supplement: No meal matrix with PPS
- Drink with placebo (Placebo Comparator): Iron-fortified drink labelled with stable iron isotope as ferrous sulfate, consumed with placebo supplement (maltodextrin).
  Interventions: Dietary Supplement: No meal matrix with placebo

INTERVENTIONS:
Dietary Supplement: Meal matrix with polyphenol supplement (PPS) — Test meal with polyphenol supplement
  Arms: Meal with polyphenol supplement (PPS)
Dietary Supplement: Meal matrix with placebo — Test meal with placebo (maltodextrin) supplement
  Arms: Meal with placebo
Dietary Supplement: No meal matrix with PPS — Test drink with polyphenol supplement
  Arms: Drink with PPS
Dietary Supplement: No meal matrix with placebo — Test drink with placebo (maltodextrin) supplement
  Arms: Drink with placebo

SUMMARY:
Genetic disorders, such as thalassemia, can lead to iron overload and severe adverse health outcomes. In iron-loading thalassemia, iron overload is due to increased iron absorption. Iron accumulates in the body organs causing widespread damage. The standard treatment is iron chelation therapy and/or periodic phlebotomy to remove iron from the body; frequency of phlebotomy or chelation therapy is dependent on how quickly body iron stores accumulate.

Polyphenolic compounds are very strong inhibitors of non-heme iron absorption, as they form insoluble complexes with ferrous iron in the gastrointestinal tract that cannot be absorbed.

The investigators have recently shown in European subjects with hereditary hemochromatosis (another iron-loading disorder) that our newly-developed natural polyphenol supplement (PPS) that is rich in polyphenols, when taken with iron-rich meals or with an iron-fortified drink, reduces iron absorption by ~40%. Decreasing non-heme iron absorption in adults with iron-loading thalassemia could potentially lead to an extension of the time period between phlebotomies or chelation therapies, and therefore an improved quality of life.

Therefore, in this stable iron isotope study, the investigators will study the effect the natural PPS on oral iron absorption from an iron-rich test meal or iron-fortified drink in Thai adults with iron-loading thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of thalassemia minor or intermedia (β-thalassemia with or without α-globin gene mutations, Hb E/β-thalassemia with or without α-globin gene mutations, or α-thalassemia Hb H disease) based on Hb electrophoresis/HPLC and/or DNA analysis from the subject's medical record.
* Hemoglobin (Hb): 7.0-13.5 g/dL for males; 7.0-12.0 for females
* Serum ferritin (SF): 300-800 ug/L for males; 200-800 ug/L for females
* Not having had a blood transfusion within 6 months prior to the study start
* Age 18-49 y, not pregnant or lactating
* Body weight <75 kg and body mass index (BMI) between 17 and 25 kg/m2
* No acute illness/infection (self-reported)
* No metabolic or gastrointestinal disorders, eating disorders or food allergy to the ingredients of the test meal (self-reported)
* No scheduled phlebotomy or blood transfusion during the study period
* The last phlebotomy will be at least 4 weeks prior to first study visit
* No intake of iron chelators 4 weeks prior to first study visit and throughout the study period
* No use of medications affecting iron absorption or metabolism during the study
* No intake of mineral/vitamin supplements 2 weeks prior to the first study visit and during the study
* No participation in any other clinical study within the last 30 days and during the study
* Expected to comply with study protocol

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Difference in fractional iron absorption (FIA) from iron-rich test meal administered with and without the polyphenol supplement (PPS). | Measured 14 days after administration of last test meal (study day 18 or 35)
  FIA from labelled test meals consumed with the PPS and consumed with the placebo will be determined based on the shift of the iron isotope ratios in whole blood.
Difference in FIA from iron-fortified test drink administered with and without the PPS. | Measured 14 days after administration of last test drink (study day 18 or 35)
  FIA from labelled test drink consumed with the PPS and consumed with the placebo will be determined based on the shift of the iron isotope ratios in whole blood.

SECONDARY OUTCOMES:
Serum ferritin (µg/L) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  to assess iron status
Soluble transferrin receptor (mg/L) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  to assess iron status
Transferrin saturation (%) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  to assess iron status
Hemoglobin (g/dL) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  to identify anemia and to determine blood volume
C-reactive protein (mg/L) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  To assess inflammation status
Alpha-1-glycoprotein (g/L), | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  To assess inflammation status
Serum hepcidin (nM) | At baseline (study day 1), midpoint (study day 18), and endpoint (study day 35)
  Major regulator of non-heme iron absorption

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD, PhD, Study Director — ETH Zurich
Locations (1):
- Mahidol University, Salaya, Thailand